CLINICAL TRIAL: NCT00247403
Title: Phase I Clinical Trial: 2DG + Stereotactic Radiosurgery (SRS) Protocol for Treatment of Intracranial Metastases
Brief Title: Safety Study of 2DG With Stereotactic Radiosurgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Pharmaceutical company no longer manufactures drug
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, John M. Buatti, Professor and Chair, Department of Radiation Oncology, University of Iowa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200506744
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Intracranial Neoplasms; Neoplasm Metastasis
Keywords: Intracranial cancer; Cancer; 2DG; 2-deoxyglucose; Intracranial metastatic cancer
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Deoxyglucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2DG (Experimental)
  Interventions: Drug: 2-deoxyglucose (2DG)

INTERVENTIONS:
Drug: 2-deoxyglucose (2DG) — Addition of 2DG to stereotactic radiosurgery. Dose escalation study.

SUMMARY:
Ionizing radiation produces cancer cell death by creating high levels of reactive oxygen species (ROS), such as superoxide and hydrogen peroxide, in irradiated cells. Cancer cells are preferentially affected by ROS. The investigators, therefore, propose that interfering with the detoxification of ROS will make radiation more toxic to cancer cells. Several cellular mechanisms exist to detoxify ROS, and glucose metabolism plays an important role in many of these mechanisms. The investigators propose that interfering with glucose metabolism will sensitize cancer cells to radiation.

The investigators' central hypothesis is that 2DG will sensitize cancer cells to ionizing radiation by inhibiting the use of glucose to detoxify reactive oxygen species produced by radiation. As an initial step to evaluate this hypothesis, the investigators have designed this phase I study.

DETAILED DESCRIPTION:
Radiosurgery is a proven treatment option for intracranial metastases. This trial is an initial effort to potentiate the therapeutic effect of single dose stereotactic radiosurgery by combining a radiation sensitizing agent, 2DG, with radiosurgery in the treatment of intracranial metastases. Our preclinical studies indicate the degree of cancer cell radiosensitization using 2DG increases with increasing radiation dose. We therefore are interested to use 2DG with radiosurgery, since this technique allows for delivery of a large single dose of radiation.

This trial seeks to determine the maximum tolerable one time dose of 2DG that can be delivered to subjects receiving stereotactic radiosurgery. We will also measure the physiologic effects of 2DG on glucose and reactive oxygen species metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Brain metastases from histologically confirmed extracranial cancer or previously confirmed intracranial carcinoma. Carcinoma must be staged using the American Joint Committee on Cancer (AJCC) staging criteria version 6.
* Morphologically well-defined tumor mass on computed tomography (CT)/magnetic resonance imaging [MRI] (largest diameter less than 40 mm) after resection.
* Intracranial mass or masses ≤ 4 cm in greatest diameter. Patients with multiple masses will be eligible if their radiosurgery treatment time is expected to last less than one hour (typically a maximum of 6 lesions).
* Standard institutional radiotherapeutic treatment is stereotactic radiosurgery delivered using bite-plate localization.
* Greater than or equal to 21 years of age. Pediatric subjects represent a minority of patients who otherwise meet the eligibility criteria. Inclusion of children in a different study would be considered if therapy is found to be effective in adults and not as part of this trial because the safety of 2DG in children has not been investigated.
* Karnofsky greater than or equal to 70% at time of screening
* Life expectancy of greater than 3 months
* Subjects must have normal organ and marrow function as defined below:

  * serum glucose < 200 mg/dl
  * hemoglobin A1C (HbA1c) < 8.5 %
* Contraceptive use in men and women of childbearing potential prior to, and for the duration of, this study. The teratogenic effects of ionizing radiation are well documented, and 2DG has the potential for teratogenic or abortifacient effects.
* Nursing of infants must be suspended during the study. There is an unknown but potential risk for adverse events in infants nursing from patients treated with 2DG, therefore breastfeeding must be discontinued for the duration of the study.
* Ability to ingest 50 ml of fluid either by mouth or feeding tube.
* Inclusion of women and minorities: Both men and women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Subjects with diabetes mellitus, elevated HbA1c or elevated blood glucose.
* Subjects requiring a headring ('halo') immobilization for standard stereotactic localization. Patients with metastases adjacent to optic chiasm, optic nerve or other radiosensitive tissue necessitating the accuracy of a headring will be excluded.
* Subjects must not be receiving any other investigational agents.
* Subjects with a history of myocardial infarction in the past year and/or dependent on beta-adrenergic blocking agents.
* Subjects with an uncontrolled seizure disorder.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the nursing mother with 2DG, breastfeeding must be discontinued while the nursing mother is treated.
* Pregnant women are excluded from this study. The teratogenic effects of ionizing radiation are well documented, and 2DG has the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative pregnancy test result immediately prior to the study and should they become pregnant or suspect that they are pregnant during the study, they must inform their treating physicians immediately.
* Inclusion of prisoners and other vulnerable populations: Prisoners and other vulnerable populations, such as children, will not be enrolled.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Safety | During treatment and 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: John M. Buatti, M.D., Principal Investigator — University of Iowa Hospitals & Clinics
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States